CLINICAL TRIAL: NCT07005492
Title: Factors Affecting Success and Survival Rates in Root Canal Retreatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Burhan Can Çanakçi, Associate Professor, Trakya University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TUTF-2023\228
Record Dates: First submitted 2025-01-13; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-01

CONDITIONS: Root Canal Therapy; Root Canal Retreatment
Keywords: root canal retreatment; non-surgical root canal treatment; survival; success
MeSH Terms: interventions — Physical Examination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radiological and clinical examination (Other): The patients were examined radiologically and clinically.
  Interventions: Diagnostic Test: radiological and clinical examination

INTERVENTIONS:
Diagnostic Test: radiological and clinical examination — Standard radiological (periapical radiography) and clinical (inspection, percussion, palpation tests etc.) examinations were performed.

SUMMARY:
The aim of this study is to evaluate the effects of pre-treatment and procedural factors on survival and success rates in teeth that underwent non-surgical root canal retreatment at Trakya University, Faculty of Dentistry between 2015-2017.

Pre-treatment factors examined:

* Age
* Gender
* Presence and size of periapical lesion
* Quality of root canal obturation

Factors examined during treatment:

* Type of restoration
* Status of restoration at recall

The null hypothesis was that these factors have no effect on survival and success rate.

DETAILED DESCRIPTION:
Patients with teeth that had undergone non-surgical recurrent root canal treatment at Trakya University, Faculty of Dentistry between 2015-2017 were invited for examination. Clinical and radiological examinations were performed on patients who agreed to participate in the study. No additional interventional procedures were performed. As a result of radiological and clinical examinations, whether the tooth was in the mouth, its clinical and radiological health, current clinical symptoms, etc. were determined.

ELIGIBILITY:
Inclusion Criterias:

* At least 18 years old at the time of treatment
* Systemically healthy (ASA 1-2)
* Acceptable obturation quality after treatment

Exclusion Criterias:

* Precense of seperated instrument before or after treatment
* Precense of perforation before or after treatment
* Apical surgery before of before or after treatment
* Immature root development
* Two adjacent teeth which required root canal treatment or treatment
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Survival rate | 78.47 ± 10.48 months after treatment
  Survival Rate:
  Survival was assessed whether the tooth was in the mouth or not. Survival was scored positive if the tooth was in the mouth, regardless of the health status of the tooth in the clinical and radiological examination at the follow-up appointment.
Success rate | 78.47 +10.48 months
  Success Rate:
  Scored as successful or unsuccessful according to the following effects according to the clinical and radiological examinations; restoration status, health of the periapical tissues, presence of swelling and/or the sinus tract.
  Success: The tooth had no clinical signs or symptoms, and the radiographs revealed complete resolution of periapical lesion Failure: The size of the periapical lesion was unchanged or increased or not completely healed, with or without clinical signs or symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Burhan Can Çanakçş, Associate professor, Study Director — Trakya University, Faculty of Dentistry, Department of Endodontics
Locations (1):
- Trakya University, Faculty of Dentistry, Edirne, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No